CLINICAL TRIAL: NCT03548298
Title: Antireflux Ablation Therapy (ARAT) With Hybrid-APC (Argon Plasma Coagulation) for GERD Treatment in Patients Without Hiatal Hernia
Brief Title: Antireflux Ablation Therapy (ARAT) for Gastroesophageal Reflux Treatment
Acronym: ARAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-2018-3601-014
Record Dates: First submitted 2018-05-23; First posted 2018-06-07 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-07

CONDITIONS: Gastro Esophageal Reflux
Keywords: GERD, Hybrid-APC, efficacy, safety; ARAT
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: Men and women with diagnosis of GERD confirmed by endoscopy or pHmetry, GERD questionnaire and that accept this new treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GERD without hiatal hernia (Experimental): Participants with GERD without hernia hiatal will receive ARAT
  Interventions: Procedure: ARAT

INTERVENTIONS:
Procedure: ARAT — After confirmation of GERD, participants will undergo to ablation with Hybrid-APC (ARAT). Participant will be admitted to hospital 24 hrs before procedure. Technique consist in ablation with hybrid-APC, submucosal injection of saline solution with methylene blue at 3-4 cm from 60-70% cardias and 1 cm esophageal. After procedure they will be kept on surveillance and will be followed-up with clinical, endoscopic, esophageal manometry and pHmetry up to 1 year after procedure.

SUMMARY:
Gastroesophageal Reflux Disease (GERD) is defined as the rise of gastric or gastroduodenal contents above the esophagogastric junction (EGJ), generating symptoms and/or esophageal lesions. It is estimated a failure to treatment with PPI(proton pump inhibitor) between 10%-40% of patients with GERD. The main disadvantages of surgical treatment include perforation (0-4%), bleeding (<1%) and pneumothorax (0-10%), the most common late complication is gastric fullness, which occurs in almost all patients, approximately 25% of patients may experience persistent dysphagia 3 months after surgery and the most worrisome late complication is the need of a new surgical intervention. The aims of treatment at EGJ is to reduce gastroesophageal reflux contents into the esophagus. Hybrid-APC with ablation of EGJ (ARAT) is a new technique with could generate a scar remodeling this region and consequently reducing reflux disease. Our objective is to evaluate the safety and efficacy of ARAT in a group of patients with GERD without hiatal hernia.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease is a condition in which there is a rise of gastroduodenal contents into the esophageal lumen, causing mucosal damage. Among treatments, medications are the most common used ones but up to 10%-40% doesn't respond to this type of treatment. Surgical treatment has been considered as the gold standard; however, with complications such as bleeding, perforation, or dysphagia after surgery. Moreover, not all patients are candidates to receive this type of treatment. Based on these data, new techniques have been explored in order to reduce morbidity, mortality and costs in the treatment of these patients.

Among different endoscopical treatments, ablation of EGJ is a new promising technique which can be used to perform a closure at this level throughout the scar secondary to hybrid-APC treatment, consequently decreasing gastroesophageal reflux. So, the aim of this study is to evaluate safety and efficacy of ARAT in a group of patients with confirmed GERD.

This is a quasi experimental study that will be conducted in a tertiary care center in Mexico city, Mexico. In an endoscopy department at the Mexican Institute of Social Security between January 2018 and July 2019. Those patients diagnosed with gastroesophageal reflux who are candidates and who accept this type of treatment will be evaluated. Patients who meet the inclusion criteria will be the definitive candidates. The risks and benefits of this type of endoscopic treatment will be explained as well as the potential scope of this endoscopic alternative. We will evaluate safety and efficacy of this new procedure.

The technique of the procedure involves ablation of the mucosa of the EGJ using Hybrid-APC (ARAT). The ablation field is initially marked with a Hybrid-APC. Subsequently, saline solution mixed with indigo-carmine is injected at the submucosa level to raise a submucosal bleb, followed by ablation of the mucosa along the lesser curvature. The approximate duration of the procedure is 40min.

Follow-up will include objective evaluation of reflux disease with: upper endoscopy, manometry, pHmetry, reflux questionnaire, and need of PPI (proton-pump inhibitor) dose quantification.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes of age with a diagnosis of GERD and who are under medical treatment and who do not wish to undergo surgical treatment
* Confirmed diagnosis of GERD in the following way:
* Positive pHmetry
* Positive endoscopy (GERD with esophagitis of any degree) or negative
* Positive symptoms questionnaire for GERD
* Manometry without evidence of esophageal motor disorder
* Total or partial response to proton pump inhibitors

Exclusion Criteria:

* Patients who do not accept the signature of the informed consent
* Patients previously treated by surgery for GERD
* Pregnant women.
* Patients with hiatal hernia greater than 3 cm or Hill type IV
* Patients with esophageal motility disorders
* Patients in whom, for any reason, any antireflux surgery or endoscopic treatment has been contraindicated.
* Patients who want to undergo surgical treatment as an initial option.
* Patients with portal hypertension and the presence of esophageal varices
* Patients with hemophilia or a haematological disorder that is difficult to control

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2016-01-10 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of ARAT with Hybrid-APC in patients with GERD without hiatal hernia | One year
  The efficacy of this treatment will be defined as: The decrease of ≥ 50 percent of the total percentage of acid exposure at 24 hrs (DeMeester Score)

SECONDARY OUTCOMES:
Safety of ARAT with hybrid-APC in patients with GERD without hiatal hernia | One Year
  We will document any adverse event presented during or after application of ARAT therapy

CONTACTS AND LOCATIONS:
Overall Officials: Oscar V Hernández Mondragón, MD, Principal Investigator — IMSS
Locations (1):
- Centro Medico Nacional Siglo XXI, Hospital de Especialidades, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mezerville Cantillo Ld, Cabas Sanchez J, Contreras F, Castellanos Garcia LF, Dondis JE, Galdamez J, Garcia-Maradiaga R, Grullon Dickson F, Jerez Gonzalez LE, Mayo DiBello M, Mejia Rivas MA, Moreno Padilla P, Sanchez Hernandez MA, Velasco SR, Vela MF, Valdovinos-Diaz MA, Remes-Troche JM. [Practice guideline of the Centroamerican and Carribean Association of Gastroenterology and Gastrointestinal Endoscopy for the management of gastroesophageal reflux disease]. Acta Gastroenterol Latinoam. 2014 Jun;44(2):138-53. No abstract available. Spanish. PMID 25199309
- [Result] Katz PO, Gerson LB, Vela MF. Guidelines for the diagnosis and management of gastroesophageal reflux disease. Am J Gastroenterol. 2013 Mar;108(3):308-28; quiz 329. doi: 10.1038/ajg.2012.444. Epub 2013 Feb 19. No abstract available. PMID 23419381
- [Result] Bolier EA, Kessing BF, Smout AJ, Bredenoord AJ. Systematic review: questionnaires for assessment of gastroesophageal reflux disease. Dis Esophagus. 2015 Feb-Mar;28(2):105-20. doi: 10.1111/dote.12163. Epub 2013 Dec 18. PMID 24344627
- [Result] Hansdotter I, Bjor O, Andreasson A, Agreus L, Hellstrom P, Forsberg A, Talley NJ, Vieth M, Wallner B. Hill classification is superior to the axial length of a hiatal hernia for assessment of the mechanical anti-reflux barrier at the gastroesophageal junction. Endosc Int Open. 2016 Mar;4(3):E311-7. doi: 10.1055/s-0042-101021. Epub 2016 Feb 10. PMID 27004249
- [Result] Villa N, Vela MF. Impedance-pH testing. Gastroenterol Clin North Am. 2013 Mar;42(1):17-26. doi: 10.1016/j.gtc.2012.11.003. PMID 23452628
- [Result] Wileman SM, McCann S, Grant AM, Krukowski ZH, Bruce J. Medical versus surgical management for gastro-oesophageal reflux disease (GORD) in adults. Cochrane Database Syst Rev. 2010 Mar 17;(3):CD003243. doi: 10.1002/14651858.CD003243.pub2. PMID 20238321
- [Result] Nabi Z, Reddy DN. Endoscopic Management of Gastroesophageal Reflux Disease: Revisited. Clin Endosc. 2016 Sep;49(5):408-416. doi: 10.5946/ce.2016.133. Epub 2016 Sep 30. PMID 27744659
- [Result] Inoue H, Ito H, Ikeda H, Sato C, Sato H, Phalanusitthepha C, Hayee B, Eleftheriadis N, Kudo SE. Anti-reflux mucosectomy for gastroesophageal reflux disease in the absence of hiatus hernia: a pilot study. Ann Gastroenterol. 2014;27(4):346-351. PMID 25330784
- [Result] Manner H, Neugebauer A, Scharpf M, Braun K, May A, Ell C, Fend F, Enderle MD. The tissue effect of argon-plasma coagulation with prior submucosal injection (Hybrid-APC) versus standard APC: A randomized ex-vivo study. United European Gastroenterol J. 2014 Oct;2(5):383-90. doi: 10.1177/2050640614544315. PMID 25360316
- [Result] Manner H, May A, Kouti I, Pech O, Vieth M, Ell C. Efficacy and safety of Hybrid-APC for the ablation of Barrett's esophagus. Surg Endosc. 2016 Apr;30(4):1364-70. doi: 10.1007/s00464-015-4336-1. Epub 2015 Jun 24. PMID 26104794
- [Derived] Hernandez Mondragon OV, Zamarripa Mottu RA, Garcia Contreras LF, Gutierrez Aguilar RA, Solorzano Pineda OM, Blanco Velasco G, Murcio Perez E. Clinical feasibility of a new antireflux ablation therapy on gastroesophageal reflux disease (with video). Gastrointest Endosc. 2020 Dec;92(6):1190-1201. doi: 10.1016/j.gie.2020.04.046. Epub 2020 Apr 25. PMID 32343977